CLINICAL TRIAL: NCT05918172
Title: Comparison of the Frequency of Ventilator-Associated Pneumonia in Intubated Patients Followed Up With Automatic Cuff Pressure Controller and Manual Cuff Pressure Controller in Pediatric Intensive Care; A Randomized Controlled Study
Brief Title: Comparison of the Frequency of Ventilator-Associated Pneumonia in Intubated Patients Followed Up With Automatic Cuff Pressure Controller and Manual Cuff Pressure Controller in Pediatric Intensive Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ayse Asik, MD, Istanbul Medeniyet University
Other Study IDs: 17334652306
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Ventilator-associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- manual group: The cuff pressure of the tracheal tube will be monitored every 8 hours in the manual group using a portable manometer. The target endotracheal tube cuff pressure will be 20 cm H2O throughout the follow-up of the patients.
  Interventions: Device: endotracheal cuff pressure manual measurement
- automatic group: The cuff pressure of the tracheal tube will be monitored continuously using a pneumatic device in the automatic group. The target endotracheal tube cuff pressure will be 20 cm H2O during the follow-up of patients.
  Interventions: Device: endotracheal cuff pressure automatic measurement

INTERVENTIONS:
Device: endotracheal cuff pressure manual measurement — The cuff pressure of the tracheal tube will be monitored every 8 hours in the manual group using a portable manometer. The target endotracheal tube cuff pressure will be 20 cm H2O during the follow-up of patients. Before starting to work, PICU nurses will be given training in recognizing and preventing VAP and using cuff pressure measuring devices. The application period will continue from the day of intubation to extubation or a maximum of 14 days. Study data forms will be filled out by PICU nurses and monitored by physicians. The research group will periodically observe PICU personnel to verify adherence to the protocol. While patients are mechanically ventilated, VIP findings will be routinely screened at each daily visit.
  Groups: manual group
Device: endotracheal cuff pressure automatic measurement — The cuff pressure of the tracheal tube will be monitored continuously using a pneumatic device in the automatic group. The target endotracheal tube cuff pressure will be 20 cm H2O during the follow-up of patients.
  Before starting to work, PICU nurses will be given training in recognizing and preventing VAP and using cuff pressure measuring devices.
  The application period will continue from the day of intubation to extubation or a maximum of 14 days Study data forms will be filled out by PICU nurses and monitored by physicians. The research group will periodically observe PICU personnel to verify adherence to the protocol. While patients are mechanically ventilated, VIP findings will be routinely screened at each daily visit.
  Groups: automatic group

SUMMARY:
Based on the hypothesis that keeping the endotracheal cuff pressure in the optimum range will reduce the incidence of vip, we aimed to compare the Manual (intermittent) measurement method with the Automatic (continuous) measurement method in reducing the incidence of vap.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VIP) is a major cause of morbidity and mortality in intensive care patients. Microaspiration of oropharyngeal and gastric secretions contaminated with bacteria is one of the important factors contributing to the formation of VIP. Under- or over-inflation of the endotracheal tube balloon (cuff) can lead to micro-aspiration, VIP development, and tracheal damage. Intermittent (manual) or continuous (automatic) control of the endotracheal tube cuff pressure has been used as a strategy for preventing VIP in recent years. There are few adult studies evaluating the effectiveness of the use of manual and automatic cuff gauges in intensive care patients in preventing the development of VIP. Our study is the first randomized controlled study in the literature to evaluate the effectiveness of two methods in preventing the development of VIP in pediatric intensive care patients.

Our study is a randomized controlled single-blind clinical study. It was planned to include patients aged between 1 month and 18 years, who required at least 48 hours of mechanical ventilation. Our exclusion criteria; intubation history in the last 14 days, airway trauma, airway anomaly, tracheotomy, mechanical ventilation for less than 48 hours and immunosuppression. It was planned to include the patients included in the study in the manual or automatic cuff gauge group using a 1:1 randomization table. In the automatic cuff meter group, it was planned to monitor the patients continuously by targeting 20 cmH20 endotracheal tube pressure. It was planned to measure the cuff pressure at 8 hour intervals for the patients in the manual cuff gauge group and to correct the deviations in the pressure. CDC criteria will be used as VIP diagnostic criteria. Patients will be monitored for the development of VIP and complications related to the endotracheal tube (such as stenosis, stridor)

ELIGIBILITY:
Inclusion Criteria:Pediatric patients aged 1 month to 18 years who required at least 48 hours of mechanical ventilation were included in the study before the 24th hour of intubation and mechanical ventilation -

Exclusion Criteria:history of intubation in the last 14 days, tracheomalacia secondary to trauma, stridor, suspected tracheal stenosis, refusal to participate in the study, presence of tracheotomy, mechanical ventilation for less than 48 hours, mechanical ventilation for more than 24 hours at PICU admission , suspected or diagnosed immunodeficiency, history of malignant disease (active or in remission), chronic pulmonary and/or heart disease, chronic other systemic diseases, and use of immunosuppressive medication (such as corticosteroids).

-

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1 month to 18 years who required at least 48 hours of mechanical ventilation in picu
Sampling Method: Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of VIP incidences | january 2022 - january 2024
  The comparison of the VIP incidence in the patients followed in the manual and automatic cuff pressure measurement groups was determined as the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- IstanbulMU, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marjanovic N, Boisson M, Asehnoune K, Foucrier A, Lasocki S, Ichai C, Leone M, Pottecher J, Lefrant JY, Falcon D, Veber B, Chabanne R, Drevet CM, Pili-Floury S, Dahyot-Fizelier C, Kerforne T, Seguin S, de Keizer J, Frasca D, Guenezan J, Mimoz O; AGATE Study Group. Continuous Pneumatic Regulation of Tracheal Cuff Pressure to Decrease Ventilator-associated Pneumonia in Trauma Patients Who Were Mechanically Ventilated: The AGATE Multicenter Randomized Controlled Study. Chest. 2021 Aug;160(2):499-508. doi: 10.1016/j.chest.2021.03.007. Epub 2021 Mar 13. PMID 33727034
- [Background] Lorente L, Lecuona M, Jimenez A, Lorenzo L, Roca I, Cabrera J, Llanos C, Mora ML. Continuous endotracheal tube cuff pressure control system protects against ventilator-associated pneumonia. Crit Care. 2014 Apr 21;18(2):R77. doi: 10.1186/cc13837. PMID 24751286
- See also: Related Info — http://www.biomedcentral.com/1471-2253/13/50